CLINICAL TRIAL: NCT05746039
Title: Feasibility of Semaglutide Therapy for Weight Loss in Advanced Lung Disease: A Pilot Study
Brief Title: Feasibility of Semaglutide in Advanced Lung Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 852967
Record Dates: First submitted 2023-02-02; First posted 2023-02-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Interstitial Lung Disease; Chronic Obstructive Pulmonary Disease; Sarcoidosis, Pulmonary; Pulmonary Hypertension
Keywords: semaglutide
MeSH Terms: conditions — Obesity; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Sarcoidosis, Pulmonary; Hypertension, Pulmonary | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Drug (semaglutide) (Experimental): Semaglutide Pen Injector 1.0 mg weekly Once weekly subcutaneous injection Other Name: Wegovy
  Interventions: Drug: Semaglutide Pen Injector

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Once weekly subcutaneous injection
  Other Names: Ozempic

SUMMARY:
The goal of this clinical trial is to learn whether semaglutide, an FDA-approved treatment for diabetes and obesity, is feasible and tolerable in patients with advanced lung disease.

The main question[s] it aims to answer are:

1. Are patients with advanced lung disease able to tolerate semaglutide therapy?
2. Are we able to titrate semaglutide therapy to a target weight?

Participants will be asked to perform pulmonary function, physical function and body composition testing, as well as a blood draw before and after 12-weeks of semaglutide therapy. While on therapy, subjects will be surveyed regarding any adverse events or side effects.

DETAILED DESCRIPTION:
This is a small open-label pilot clinical trial of semaglutide in adults (age 18 or older, n=8) with obesity (BMI≥30 kg/m2), and chronic advanced lung disease (interstitial lung disease, sarcoidosis, chronic obstructive pulmonary disease, or pulmonary hypertension requiring supplemental oxygen on exertion). This study will evaluate medication adherence and side effects to determine semaglutide tolerability. Markers of physical function and pulmonary function will be evaluated before therapy and after 12 weeks of therapy to determine the effect of semaglutide on function. Measures of fat and muscle, will be performed before therapy and after 12 weeks of therapy to evaluate how semaglutide alters body composition in this population. Study participants will be monitored for 12 weeks while receiving semaglutide therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following lung diseases: interstitial lung disease, sarcoidosis, chronic obstructive pulmonary disease, or pulmonary hypertension
* Age > 18
* BMI > 30 kg/m2
* Requires supplemental oxygen on exertion
* Stable treatment regimen X 90 days
* Use of disease-modifying therapy

Exclusion Criteria:

* Diabetes
* Pregnant or Breastfeeding
* Recent weight loss
* Recent or chronic GI complaints
* History of gastroparesis
* History of scleroderma
* Hospitalized at time of evaluation
* Use of weight loss medication in last 90 days
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia (type 2)
* Uncontrolled thyroid disease
* History of acute/chronic pancreatitis
* Prior suicide attempt
* Suicidal ideation in last 90 days
* Presence of a pacemaker or defibrillator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Tolerability | 12 weeks
  The proportion of participants who either reach a target semaglutide dose of 1.0 mg/week or who achieve target weight.

SECONDARY OUTCOMES:
Body composition | Baseline to 12 weeks
  Change in percent body fat
Body composition | Baseline to 12 weeks
  Change in skeletal muscle index
Body composition | Baseline to 12 weeks
  Change in weight
Lung function | Baseline to 12 weeks
  Change in forced vital capacity
Lung function | Baseline to 12 weeks
  Change in forced expiratory volume in 1 second
Lung function | Baseline to 12 weeks
  Change in diffusion capacity
Physical function | Baseline to 12 weeks
  Change in frailty as measured by the Short Physical Performance Battery
Physical function | Baseline to 12 weeks
  Change in six-minute walk distance
Markers of adiposity and insulin resistance | Baseline to 12 weeks
  Change in c-reactive protein
Markers of adiposity and insulin resistance | Baseline to 12 weeks
  Change in glycosylated hemoglobin
Markers of adiposity and insulin resistance | Baseline to 12 weeks
  Change in free fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Michaela R Anderson, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No